CLINICAL TRIAL: NCT00242138
Title: A Cross-Sectional Study of Erectile Dysfunction in Patients With Locally Advanced Prostate Cancer Who Have Undergone Radiotherapy and Prolonged Pharmacological Androgen Ablation
Brief Title: Erectile Dysfunction/Prostate/RT/Androgen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: UHN REB 01-0552-C
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Behavioral: Erectile Dysfunction

SUMMARY:
The optimal duration of hormonal therapy is yet to be determined in the treatment of locally advanced carcinoma of the prostate. The RTOG performed a trial of 4 months of neoadjuvant and concurrent hormones(consisting of Goserelin and Flutamide) compared to radiation alone, and found that there was an improvement in local control and progression-free survival, but no improvement in overall survival. The EORTC performed a similar trial, but used Goserelin alone for a period of 3 years. This trial showed an improvement in local control, disease-free survival, and in contrast to the RTOG trial, an improvement in overall survival.

The rate of erectile dysfunction in men who receive a prolonged period of Gosereline (i.e. 2 yrs) is not known, but suspected according to expert opinion, to be significantly higher than a shorter course of hormonal ablation. Therefore the price of of a survival advantage in locally advanced prostate cancer maybe at a cost of increased rates of erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical stage T1-T4 carcinoma of the prostate
* Must have undergone radical radiation and at least 2 years of Pharmacological androgen ablation.Pharmacological androgen ablation may include: LHRH-agonists with or without Non-steroidal androgen ablation, Steroidal Anti-androgens, Progestational agents, and Cypoterone (Androcur).
* Must be currently 6 months or more after their last injection of LHRH-agonists if it was being given every 3 months or 4 months or more after their last injection, if it was being given monthly. If the patient was on oral androgen ablation agent, they must be off this medication for a period of at least 4 months.
* currently off hormonal therapy
* Able to sign the consent form and fill out questionnaire used in the study.

Exclusion Criteria:

* No patients who have been treated, or are currently being treated with Bicalutamide
* no previous orchidectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2000-03; Study Completion 2004-04

PRIMARY OUTCOMES:
This study is designed to address absolute incidence of erectile dysfunction, as measured by the International index of Erectile function.

SECONDARY OUTCOMES:
This study is designed to address the effects of erectile dysfunction persist one year after the initial assessment of erectile dysfunction,as measured by the International index of Erectile function.

CONTACTS AND LOCATIONS:
Overall Officials: Padraig Warde, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network Princess Margaret Hospital, Toronto, Ontario, Canada